CLINICAL TRIAL: NCT03693521
Title: Does Measurement of Handgrip Strength Affect Physical Activity Level for Patients With Diabetes Type 2? A Randomized Controlled Trial
Brief Title: Effects of Measurement of Handgrip Strength on Physical Activity Level for Patients With Diabetes Type 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Collaborators: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VGFOUREG-751161
Record Dates: First submitted 2018-08-24; First posted 2018-10-03 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Diabetes Mellitus, Type 2; Physical Activity; Muscular Weakness
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Muscle Weakness | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Standard care at yearly check-up by diabetes-nurse in primary care. Handgrip strength measurement bilaterally. Measurement of physical activity level.
  Interventions: Device: Handgrip strength measurement; Other: Standard care
- Control group (Active Comparator): Standard care at yearly check-up by diabetes-nurse in primary care. Measurement of physical activity level.
  Interventions: Other: Standard care

INTERVENTIONS:
Device: Handgrip strength measurement — Measurement of handgrip strength with Jamar hand-held dynamometer as a complement to standard care of patients with diabetes type 2 by diabetes-nurses.
  Arms: Intervention group
Other: Standard care — Standard care of patients with diabetes type 2 by diabetes-nurses.

SUMMARY:
Background: It is recommended that patients with diabetes type 2 keep themselves physically active and it is known that good muscular strength has a positive effect on these patients.

Aim: To determine whether physical activity level increases and whether other risk factors for cardiovascular disease are positively affected by including measurement of handgrip strength as part of the regular care program for patients with diabetes type 2 in primary care.

Method: Patients with diabetes type 2 who go to regular check-ups by participating diabetes-nurses in primary care are randomized to either intervention or control group. In the intervention group, handgrip strength is measured in addition to standard care. the control group receives standard care at inclusion. Handgrip strength is measured in both groups at 1 year follow-up. Physical activity level is measured in both groups at inclusion and 1 year follow-up with a questionnaire. Measurement of other risk factors for cardiovascular morbidity are measured at both inclusion and follow-up in both groups as dictated by standard care routines.

Expected results: Measurement of handgrip strength can give health care personnel greater possibilities to identify those patients with diabetes type 2 who need to increase their activity level and to give them more concrete support. It is possible that the attention given to handgrip strength and physical activity may motivate patients to increase their activity level, become stronger and eventually reduce other risk factors for cardiovascular morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes type 2 who go to regular check-ups with participating diabetes-nurses at primary health care centres in Region Västra Götaland, Sweden.

Exclusion Criteria:

* No gender, age or language restrictions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 334 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Change in physical activity level | Change from baseline at 1 year.
  Two questions evaluating frequency and intensity of physical activity according to recommendations by the American College of Sports Medicine and the American Heart Association.

SECONDARY OUTCOMES:
Change in handgrip strength | Change from baseline at 1 year.
  Handgrip strength in kg measured with Jamar hand dynamometer
Change in HbA1c | Change from baseline at 1 year.
  Blood test. HbA1c level measured in mmol/mol
Change in waist circumference | Change from baseline at 1 year.
  Waist circumference in cm measured with tape measure while standing
Physical Activity on Prescription | Change from baseline at 1 year.
  Total number of prescriptions for physical activity issued by participating diabetes-nurses. Differences measured between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Margareta Hellgren, PhD, Study Director — Närhälsan; Maria EH Larsson, PhD, Study Director — Närhälsan
Locations (7):
- Sweden (7):
  - Närhälsan Angered vårdcentral, Angered
  - Närhälsan Biskopsgården vårdcentral, Gothenburg
  - Närhälsan Brämaregården vårdcentral, Gothenburg
  - Närhälsan Gamlestaden vårdcentral, Gothenburg
  - Närhälsan Kärra vårdcentral, Gothenburg
  - Närhälsan Tuve vårdcentral, Gothenburg
  - Närhälsan Stenungsund vårdcentral, Stenungsund

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bornhoft L, Bernhardsson S, Nordeman L, Grimby-Ekman A, Dottori M, Larsson MEH. Monitoring handgrip strength to motivate lifestyle choices for patients with diabetes type 2 - a pragmatic randomised controlled trial. Scand J Prim Health Care. 2024 Dec;42(4):617-632. doi: 10.1080/02813432.2024.2373298. Epub 2024 Jul 4. PMID 38963325